CLINICAL TRIAL: NCT02139865
Title: The Effects of Resistance Training Intensity on Muscular Hypertrophy and Strength in Young, Resistance Trained Men
Brief Title: The Effects of Lifting Light or Heavy Weights on Muscle Growth and Strength in Trained Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB 14-333
Record Dates: First submitted 2014-04-07; First posted 2014-05-15 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2016-03

CONDITIONS: Skeletal Muscle Hypertrophy; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30% (Experimental): Training at 30% 1RM
  Interventions: Behavioral: 30% 1RM
- 80% (Experimental): Training at 80% 1RM
  Interventions: Behavioral: 80% 1RM

INTERVENTIONS:
Behavioral: 30% 1RM — Participant exercises using a protocol tailored at 30% of their 1RM
  Arms: 30%
Behavioral: 80% 1RM — Participant exercises using a protocol tailored at 80% of their 1RM
  Arms: 80%

SUMMARY:
When practicing weightlifting regularly the body makes new proteins within the muscle.

These new proteins can increase the size of the cells within the muscle to make them larger, a process called hypertrophy. The common convention surrounding gains in skeletal muscle size and strength is that heavy weights are needed. In contrast, lifting lighter weights are thought to be required to induce muscular endurance and not to promote growth. However, it has previously been shown in untrained men that lifting lighter weights results in similar gains in muscle mass and strength as lifting heavier weights. The purpose of this study is to examine how performing resistance training of different intensities (light or heavy weights) affects the degree of muscle growth and strength gain in individuals who are already resistance training.

This information will be valuable when designing exercise protocols for increasing muscle size and strength at all ages, or in individuals returning from injury, as a way to stimulate muscle growth and promote strength gains without the need to lift heavy weights.

DETAILED DESCRIPTION:
Patients will visit the laboratory of Dr. Stuart Phillips at the Ivor Wynne Centre (IWC) at McMaster University for 14 weeks for a number of tests and exercise sessions.

Each visit will be as follows:

Visit 1:

Upon obtaining consent, eligible participants will complete a medical screening questionnaire to determine their readiness to perform exercise as well as a filling out a form to determine subject characteristics. Participants will begin collecting data for their first 3-day diet record. They will record their diet (2 weekdays and a weekend day) again at 6 weeks (mid-protocol) and at 12 weeks of the study.

Visit 2:

Participants will report the lab between 08.00 and 10.00 h to undergo body composition scans including BodPod (to assess fat mass), bioelectrical impedance (BIA - to assess your total body water content), and Dual-energy x-ray- Absorptiometry (DXA- to determine bone mineral content). All tests will be performed in the post-absorptive state (12 hours). Participants will also have a familiarization with the lab and exercise equipment to determine preliminary resistance training (RT) loads.

Visit 4:

Participants will report to the lab to determine their one-repetition-maximum on the leg press, leg extension, bench press and shoulder press. This will be done by having participants attempt a weight based on their familiarization session; if they can complete this weight though a full range of motion with good form, they will rest 3-5 min and then attempt a higher weight until their 1RM is reached.

Visit 5:

Participants will report to the lab in the post-absorptive state (12 hours) for a resting muscle biopsy from the muscle on the outside of their thigh.

Visits 6: Participants will be randomly assigned to one of two exercise intensity treatment groups: ~30% of 1RM (which equates to ~20-25 repetitions per set) for 3 sets to failure (25 subjects) or 80% of 1RM for 3 sets to failure (another 25 subjects). All sets will have 60 seconds of rest in between. On two occasions (one at the beginning of the study another at the end), participants will return to the lab in the post-absorptive state and a catheter (plastic tube with a small needle) will be inserted into a vein in your arm. A resting blood sample will be taken. Upon completion of their first exercise session, subsequent blood samples will be taken at 15 minutes, 30 minutes 60 minutes to determines an acute time course of the changes in blood metabolites and hormones.

Visit 7-54:

Participants will attend supervised exercise sessions 4 times per week (Monday, Tuesday, Thursday and Friday) alternating lower body and upper body focused sessions for 12 weeks. Participants in the 30% (LOW) group will perform approximately 20-25 repetitions per set while participants in the 80% (HIGH) group will perform approximately 8-12 repetitions per set. Immediately following each resistance training session as well as prior to sleep, participants will consume 30g of whey protein. 1RM testing will be repeated every three weeks throughout the protocol and will be conducted prior to beginning the last of every 12 training sessions. Prior to completing their final training session (session number 48) participants will again arrive to the lab in the post-absorptive state for blood sampling procedure as described previously.

Visit 55:

Participants will arrive in the post absorptive (fasted) state 48 hours following their last training session. They will undergo a final BodPod, DEXA and BIA scan to determine body composition as well as a final resting biopsy of the vastus lateralis muscle.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-30 years old
* Non-obese (Body mass index less than 30 kg/m2)
* Non-smoker
* Healthy based on questionnaire responses (see exclusion criteria)
* Resistance trained (Resistance training > 2 times per week for 2 years, minimum 1 lower body exercise session per week)

Exclusion Criteria:

* Allergies to milk proteins (whey or casein)
* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through medical history screening questionnaires
* Arthritic conditions
* Individuals who consume any analgesic or anti-inflammatory drug(s), prescription or non- prescription, chronically will be excluded
* A history of neuromuscular problems
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Muscle Volume | 0 weeks (baseline) and 12 weeks
  Change from baseline at 12 weeks Measured via 4 compartment model

SECONDARY OUTCOMES:
Gene expression | 0 weeks (baseline) and 12 weeks
  Change from baseline at 12 weeks . Gene expression for proteins involved in muscle protein synthesis measured from muscle biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario

REFERENCES:
- [Result] Morton RW, Oikawa SY, Wavell CG, Mazara N, McGlory C, Quadrilatero J, Baechler BL, Baker SK, Phillips SM. Neither load nor systemic hormones determine resistance training-mediated hypertrophy or strength gains in resistance-trained young men. J Appl Physiol (1985). 2016 Jul 1;121(1):129-38. doi: 10.1152/japplphysiol.00154.2016. Epub 2016 May 12. PMID 27174923